CLINICAL TRIAL: NCT06199609
Title: Changes in Cardiac Structure and Function in Patients With End-stage Renal Disease After Establishment of Autologous Arteriovenous Fistula
Brief Title: Changes in Cardiac Structure and Function After Establishment of Autologous Arteriovenous Fistula
Status: Completed | Type: Observational
Sponsor: Haiyan Wang (Other)
Responsible Party: Sponsor-Investigator, Haiyan Wang, Director of Cardiac Ultrasound, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023（130）
Record Dates: First submitted 2023-12-11; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: End Stage Renal Disease; Arteriovenous Fistula
Keywords: ESRD; AVF; MHD; AF; Echocardiogram
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AVF group and TCC group: AVF and TCC are two different hemodialysis pathways
  Interventions: Procedure: Hemodialysis pathway
- Before AVF establishment and After AVF establishment: Evaluate and analyze the changes in cardiac structure and function before and after the establishment of AVF;
  Interventions: Procedure: AVF
- Left atrial enlargement group and Left atrial normal group: Patients in the AVF group are divided into a left atrial enlargement group and a left atrial normal group based on whether the left atrium has expanded after the establishment of AVF
  Interventions: Procedure: AVF
- Atrial fibrillation group and Non atrial fibrillation group: Divide AVF group patients into atrial fibrillation group and non atrial fibrillation group based on whether new atrial fibrillation occurs after AVF establishment
  Interventions: Procedure: AVF

INTERVENTIONS:
Procedure: Hemodialysis pathway — AVF and TCC are two different vascular pathways for hemodialysis
  Groups: AVF group and TCC group
Procedure: AVF — Left atrial changes caused by AVF establishment
  Groups: Before AVF establishment and After AVF establishment; Left atrial enlargement group and Left atrial normal group
Procedure: AVF — New onset atrial fibrillation caused by AVF establishment
  Groups: Atrial fibrillation group and Non atrial fibrillation group

SUMMARY:
This study is a retrospective cohort study aimed at evaluating the impact of autologous arteriovenous fistula (AVF) on the heart, especially the left atrial structure, in patients with end-stage renal disease (ESRD) through a retrospective cohort study. The aim is to further clarify the relationship between the establishment of AVF and the occurrence of atrial fibrillation, and provide a theoretical basis for exploring the relevant mechanisms of AVF induced atrial fibrillation in the future.

DETAILED DESCRIPTION:
1. Retrospective collection of ESRD patients who visited the Department of Nephrology at the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital, Shandong Province) from January 2014 to December 2022 for hemodialysis using AVF and tunnel cuffed catheter (TCC) with a tunnel and polyester sheath. Follow up comparison of the incidence of atrial fibrillation between the two groups;
2. Collect general clinical data (gender, age, primary disease, history, etc.), echocardiography (atrioventricular diameter, wall thickness, left ventricular ejection fraction, pulmonary artery pressure, etc.), and biochemical indicators (albumin, total bilirubin, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, blood creatinine, blood calcium, blood phosphorus, hemoglobin, etc.) of AVF patients, Analyze the changes in the structure of the heart, especially the left atrium, before and after the establishment of AVF, and use binary logistic regression to analyze the risk factors for new onset atrial fibrillation after AVF surgery;
3. According to whether new atrial fibrillation occurred after AVF surgery, patients were divided into atrial fibrillation group and non atrial fibrillation group. The occurrence of adverse clinical outcomes was followed up, and the Kaplan Meier survival curve was used to analyze the impact of atrial fibrillation on patient adverse clinical outcomes. Cox regression analysis was used to explore independent risk factors for adverse clinical outcomes.

Follow up: Follow up will be conducted by a dedicated doctor from the establishment of AVF to August 31, 2023. The main endpoint events are defined as all-cause death and cardiogenic death, while the secondary endpoint events are readmission due to heart failure and stroke; During the follow-up period, patients who underwent kidney transplantation, changed dialysis methods, and did not experience endpoint events at the end of the follow-up were defined as missing data.

ELIGIBILITY:
Inclusion Criteria:

* ① Meets the diagnostic criteria for chronic kidney disease; ② Age ≥ 18 years old; ③ Regular dialysis patients; ④ Using AVF or TCC as the sole vascular pathway.

Exclusion Criteria:

* ① Irregular dialysis patients; ② High output states such as hyperthyroidism; ③ Basic heart diseases (cardiomyopathy, severe valvular disease, intracardiac shunting, constrictive pericarditis, post heart transplant, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients who underwent hemodialysis using AVF and Tunnel Cuffed Catheter (TCC) with a polyester sleeve in the Department of Nephrology at the First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital, Shandong Province) from January 2014 to December 2022.
  The AVF group patients included in the analysis are required to undergo echocardiography examination within 3 months before and after the establishment of AVF, in order to conduct long-term and longitudinal evaluation of the cardiac structure and function of MHD patients.
Sampling Method: Non-Probability Sample
Enrollment: 2027 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence rate of atrial fibrillation | Completed through follow-up, with an average of 4 years
  Follow up comparison of the incidence of atrial fibrillation between the AVF group and the TCC group；Comparison of the incidence of atrial fibrillation before and after AVF establishment
Changes in left atrial size (anterior posterior diameter) after AVF establishment | Completed through follow-up, with an average of 2 years
  Collect echocardiography data before and after AVF establishment to compare changes in the left atrium before and after establishment
Comparison of the incidence of clinical outcomes between the atrial fibrillation group and the non atrial fibrillation group | Completed through follow-up, with an average of 2 years
  Follow up comparison of clinical outcomes between the atrial fibrillation group and the non atrial fibrillation group, and Cox regression analysis of risk factors

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Derived] Song W, Wu L, Sun C, Kong X, Wang H. New-onset atrial fibrillation following arteriovenous fistula increases adverse clinical events in dialysis patients with end-stage renal disease. Front Cardiovasc Med. 2024 Apr 12;11:1386304. doi: 10.3389/fcvm.2024.1386304. eCollection 2024. PMID 38682103